CLINICAL TRIAL: NCT02507180
Title: Safely Ruling Out Deep Vein Thrombosis in Pregnancy With the LEFt Clinical Decision Rule and D-Dimer: the LEaD Study. A Prospective Cohort Study.
Brief Title: Safely Ruling Out Deep Vein Thrombosis in Pregnancy With the LEFt Clinical Decision Rule and D-Dimer
Acronym: LEaD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University Hospital, Geneva (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20150546-01H
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy; Deep Vein Thrombosis
Keywords: Clinical Decision Rule; Ultrasound; Suspected Deep Vein Thrombosis; D-Dimer; LEFt
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At presentation, a blood sample will be collected for clinical D-dimer tested in real time and a sample will be collected and the plasma will be frozen for analysis at the end of study using Vidas D-dimer on all patient samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with suspected DVT: Pregnant women presenting with suspected DVT will have the LEFt clinical decision rule applied by the attending physician and will have a clinical D-dimer test done.
  Interventions: Other: LEFt clinical decision rule

INTERVENTIONS:
Other: LEFt clinical decision rule — The LEFt rule
  Predictor Points Left leg symptoms +1 Extremity swelling (≥ 2 cm difference in calf circumference +1 First trimester symptom onset +1
  Clinical probability Unlikely: 0 or 1 point Likely: > 1 point

SUMMARY:
This is prospective cohort study in pregnant women who present with signs and symptoms of possible deep vein thrombosis (DVT). All patients will have the same method of assessment of their DVT symptoms (the LEFt clinical decision rule will be applied and D-dimer test will be done) to determine if a compression ultrasound is required. All patients will be followed for a period of 3 months.

DETAILED DESCRIPTION:
VTE is a leading cause of maternal death in the developed world. Suspected DVT in pregnancy is a common clinical problem faced by clinicians daily. The only validated method to exclude DVT in pregnancy requires leg vein CUS imaging. This imaging modality is costly and has limited availability (only available in radiology departments and, usually, only during weekday daytime hours) often necessitating referral to the emergency room for initiation of heparin injections until leg vein CUS can be obtained. A simple and seemingly powerful clinical decision rule (LEFt) and a simple blood test (D-dimer) may be promising to exclude DVT in pregnancy without the need for diagnostic imaging. Validating the safety of a simple, non-invasive, widely available approach to suspected DVT in pregnancy would be an important advance in maternal health.

A prospective cohort diagnostic management study in pregnant women with suspected DVT, with three-month follow-up for symptomatic VTE will take place in multiple centres throughout Canada and Europe.

After obtaining informed consent, all patient will have the LEFt clinical decision rule applied by the attending physician and will have D-Dimer testing (D-Dimer results of test performed within 24 hours will be accepted and do not need to be repeated).

Patients with an "unlikely" LEFt score of 0 or 1 point and a negative D-dimer will not undergo diagnostic imaging.

Patients with either a "likely" LEFt score of 2 or 3 points or a positive D-dimer will undergo either a single complete leg vein compression ultrasound (CCUS) (Day 1) or a serial proximal leg vein (CUS) (Day 1 and Day 7).

All patients will be followed for 3 months for symptomatic VTE.

ELIGIBILITY:
Inclusion Criteria:

1. Unselected pregnant women (as self-reported by patient and/or previously documented positive beta hCG on urine or serum pregnancy tests) with
2. Suspected acute symptomatic deep vein thrombosis, defined as:

   1. New leg swelling or edema with onset in the last month or,
   2. New leg pain (buttock, groin, thigh or calf) with onset in the last month.

Exclusion Criteria:

1. Below the age of legal consent in jurisdiction of residence (18 years old for Quebec and 16 years old for rest of Canada)
2. Baseline imaging (imaging done after a minimum of 3 months of treatment for prior proximal DVT) not available if suspected recurrence in the same leg as prior
3. Unable or unwilling to provide informed consent
4. Concomitant symptoms of suspected pulmonary embolism (chest pain or shortness of breath or syncope/pre-syncope or unexplained tachycardia)
5. Therapeutic anticoagulant more than 48 hours.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unselected pregnant women presenting with suspected deep vein thrombosis
Sampling Method: Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of VTE diagnosed in patients deemed DVT "unlikely" | 3 months after presentation
  The primary outcome will be the number of VTE (distal or proximal DVT, sub-segmental or greater pulmonary embolism (PE), death attributable to VTE) documented during the three-month follow-up in those patients left untreated for DVT on the basis of the study's initial diagnostic management (see Figure 2) i.e. not doing CUS on patients with an "unlikely" LEFt score (0 or 1 points) and a negative D-dimer

SECONDARY OUTCOMES:
Number of VTE diagnosed in all patients | 3 months after presentation
  The number of major VTE events (any proximal DVT, segmental or greater PE, death attributable to VTE) documented during the 3-month follow-up in all patients. Some clinicians may not treat distal DVT or sub-segmental PE in pregnancy, instead following these patients with serial US imaging, and hence may prefer to focus on this outcome that excludes distal DVT and sub-segmental PE.
Proportion of women requiring CUS | Baseline
  The proportion of women requiring CUS using the study's diagnostic strategy (i.e. no imaging in patients with an "unlikely" LEFt score (0 or 1 points) and a negative D-dimer). We anticipate that an important proportion (>40%) of women will be able to avoid the need for CUS imaging based on safely excluding DVT on the basis of an "unlikely" LEFt (0 or 1) and a negative D-dimer. However, if this proportion is very low (<5%) this may argue against the widespread adoption of our proposed diagnostic management strategy even if it proves to be safe.
Average number of CUS in pregnant women with suspected DVT | 7 days from initial presentation
  The mean number of ultrasounds per patient with suspected DVT. In the study by Chan, validating serial CUS in pregnancy, the mean number of US per patient was 2.8630. We anticipate that we will be able to reduce this by >40% with our diagnostic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD, Principal Investigator — Ottawa Hospital Research Institute; Marc Righini, MD, Principal Investigator — Hopitaux Universitaires de Geneve
Locations (12):
- Intermountain Healthcare, Inc., Murray, Utah, United States
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Medical Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Leiden University Medical Center, Leiden, Netherlands
- Hopitaux Universitaires de Geneve, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided